CLINICAL TRIAL: NCT06039657
Title: Effectiveness of Scientific Exercise Approach to Scoliosis in Adolescents With Mild Idiopathic Scoliosis
Brief Title: Effectiveness of Scientific Exercise Approach to Scoliosis in Mild Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gözde Yagci (Gür), Assoc. Prof, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO16/82
Record Dates: First submitted 2023-09-06; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Scoliosis Idiopathic; Exercise; Quality of Life; Treatment
Keywords: scoliosis; exercise therapy; quality of life; physical appearance
MeSH Terms: conditions — Motor Activity; Scoliosis | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SEAS group (Experimental): The SEAS therapy program comprised a one-year supervised exercise regimen. Supervised sessions were scheduled weekly for the initial month, bi-weekly for the second month, and monthly from the third to the sixth month. Thereafter, sessions were held bimonthly, each lasting one hour. Home exercises were designed to encompass 10-12 distinct exercises, with an approximate duration of 40-45 minutes per session
  Interventions: Other: SEAS training
- Standard Care Group (Active Comparator): Standard care program aimed to provide patients with basic postural education and exercises in a single session, followed by one year of observation to ensure standard care.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: SEAS training — Patients who opted to participate in the SEAS group underwent SEAS therapy. The SEAS therapy program initially comrised patient education and active self-correction. Subsequently, stabilization of active self correction was tried to be performed through various functional activities. These activities were selected from everyday life examples, with increasing levels of difficulty over time. With SEAS exercises, the activation of self-correction was aimed to be increased through various activities in sitting, standing and walking conditions, with the goal of correcting scoliosis in this way
  Arms: SEAS group
Other: Standard Care — Patients who declined or were unable to participate in outpatient exercise programs received standard care. Standard care included exercises for postural re-education, traditional strengthening and stretching exercises for one session, followed by observation for one year.
  Arms: Standard Care Group

SUMMARY:
İdiopathic scoliosis is a three dimensional deformity with lateral deviation and rotation of the spine. In idiopathic scoliosis, scoliosis-specific exercises are utilized as a primary treatment for moderate curves and as a supportive measure alongside bracing for more severe curves. SEAS, which stands for Scientific Exercises Approach to Scoliosis, refers to a treatment approach developed as a scientific exercise methodology for scoliosis. This approach aims to provide scoliosis-specific exercises and techniques to manage and potentially improve the condition. This study aims to investigate the effectiveness of SEAS as a conservative treatment approach for mild AIS.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) constitutes a multifaceted distortion involving three-dimensional structural curvature of the spine, accompanied by biomechanical alterations that advance gradually, exerting an adverse influence on the quality of life related to health in individuals ranging from 10 to 18 years of age. In idiopathic scoliosis, curvatures ranging from 10 to 25 degrees are categorized as mild, while curvatures between 25 and 45 degrees are considered moderate, and those exceeding 45 degrees are classified as severe. For mild scoliosis, scoliosis specific exercises are the main treatment method. SEAS (Scientific Exercises Approach to Scoliosis), a specific type of scoliosis specific exercise program, focuses on using scientific principles to address the unique needs of individuals with scoliosis. It aims to improve posture, spinal alignment, and muscle balance through tailored exercises. SEAS exercises involve three-dimensional spinal correction and are designed to enhance neuromuscular control and proprioception in this corrective position. The available research regarding SEAS in adolescent idiopathic scoliosis (AIS) is somewhat limited both in terms of quantity and scope, underscoring the necessity for more comprehensive investigations. Drawing from the existing literature landscape and the identified gaps, our hypothesis centers on the notion that the incorporation of SEAS is poised to yield noteworthy enhancements across various dimensions of AIS. Consequently, the primary objective of this study was to assess the efficacy of SEAS training in ameliorating parameters such as Cobb angle, axial trunk rotation, bodily aesthetics, and health-related quality of life in individuals diagnosed with mild AIS. Patients in this study were treated using two different protocols based on a shared decision-making model. Patients and their families were informed about the pathology, history and progression risk of idiopathic scoliosis, as well as the exercise options and expected outcomes. Consequently, every patient along with their parents comprehensively grasped the significance of scoliosis-specific exercises in proactively rectifying and maintaining their spinal alignment throughout diverse functional activities. Patients who choose for exercise treatment underwent SEAS therapy, while those who declined or were unable to participate in outpatient exercise programs received standard care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Adolescent Idiopathic Scoliosis (AIS).
* A Cobb angle measurement falling within the range of 12° to 25°.
* Patients considered for the study were required to be within the age range of 10 to 16 years old.
* have a Risser score ranging from 0 to 4.

Exclusion Criteria:

* Patients with a history of prior spine treatment, including surgery or conservative treatment
* Patients with a history of traumatic spinal injury
* Individuals with rheumatologic disorders, which affect the joints and connective tissues
* Patients with systemic disorders, which affect multiple organ systems in the body
* Those with neurologic disorders, impacting the nervous system
* Individuals with any other musculoskeletal disorders

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Cobb angle | Measurements were performed at baseline and at the end of the one-year treatment period.
  The Cobb angle was used to quantify the degree of spinal curvature in scoliosis, determined by the angle formed by lines drawn along the endplates of the vertebrae at the curve's apex and endpoints

SECONDARY OUTCOMES:
Axial trunk rotation | Measurements were performed at baseline and at the end of the one-year treatment period.
  Axial trunk rotation measurement in the Adams test was used to the assessment of the degree of rotation of the patient's trunk while they bend forward at the waist with their arms extended downward, helping to identify any asymmetry or abnormal spinal curvature associated with scoliosis.
Spinal Appearance Questionnaire (SAQ) | Measurements were performed at baseline and at the end of the one-year treatment period.
  The Spinal Appearance Questionnaire was used as a self-reporting assessment tool used in the evaluation of individuals with spinal deformities, particularly scoliosis. It consists of a series of questions or statements designed to gather information about the patient's perception of their spinal appearance, including factors like posture, symmetry, and body image, to help in treatment planning and assessing the impact of spinal deformities on their quality of life.
Scoliosis Research Questionnaire-22 (SRS-22) | Measurements were performed at baseline and at the end of the one-year treatment period.
  SRS-22 was used in the evaluation of patients with scoliosis or spinal deformities. It assesses the patient's health-related quality of life and function through a series of questions related to pain, function, self-image, and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Halil Gokhan Demirkiran, Prof, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Samanpazari, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Negrini S, Donzelli S, Aulisa AG, Czaprowski D, Schreiber S, de Mauroy JC, Diers H, Grivas TB, Knott P, Kotwicki T, Lebel A, Marti C, Maruyama T, O'Brien J, Price N, Parent E, Rigo M, Romano M, Stikeleather L, Wynne J, Zaina F. 2016 SOSORT guidelines: orthopaedic and rehabilitation treatment of idiopathic scoliosis during growth. Scoliosis Spinal Disord. 2018 Jan 10;13:3. doi: 10.1186/s13013-017-0145-8. eCollection 2018. PMID 29435499
- [Background] Weinstein SL. The Natural History of Adolescent Idiopathic Scoliosis. J Pediatr Orthop. 2019 Jul;39(Issue 6, Supplement 1 Suppl 1):S44-S46. doi: 10.1097/BPO.0000000000001350. PMID 31169647
- [Background] Gamiz-Bermudez F, Obrero-Gaitan E, Zagalaz-Anula N, Lomas-Vega R. Corrective exercise-based therapy for adolescent idiopathic scoliosis: Systematic review and meta-analysis. Clin Rehabil. 2022 May;36(5):597-608. doi: 10.1177/02692155211070452. Epub 2021 Dec 28. PMID 34962437
- [Background] Berdishevsky H, Lebel VA, Bettany-Saltikov J, Rigo M, Lebel A, Hennes A, Romano M, Bialek M, M'hango A, Betts T, de Mauroy JC, Durmala J. Physiotherapy scoliosis-specific exercises - a comprehensive review of seven major schools. Scoliosis Spinal Disord. 2016 Aug 4;11:20. doi: 10.1186/s13013-016-0076-9. eCollection 2016. PMID 27525315
- [Background] Romano M, Negrini A, Parzini S, Tavernaro M, Zaina F, Donzelli S, Negrini S. SEAS (Scientific Exercises Approach to Scoliosis): a modern and effective evidence based approach to physiotherapic specific scoliosis exercises. Scoliosis. 2015 Feb 5;10:3. doi: 10.1186/s13013-014-0027-2. eCollection 2015. PMID 25729406
- [Background] Sanders JO, Harrast JJ, Kuklo TR, Polly DW, Bridwell KH, Diab M, Dormans JP, Drummond DS, Emans JB, Johnston CE 2nd, Lenke LG, McCarthy RE, Newton PO, Richards BS, Sucato DJ; Spinal Deformity Study Group. The Spinal Appearance Questionnaire: results of reliability, validity, and responsiveness testing in patients with idiopathic scoliosis. Spine (Phila Pa 1976). 2007 Nov 15;32(24):2719-22. doi: 10.1097/BRS.0b013e31815a5959. PMID 18007251
- [Background] Asher M, Min Lai S, Burton D, Manna B. Discrimination validity of the scoliosis research society-22 patient questionnaire: relationship to idiopathic scoliosis curve pattern and curve size. Spine (Phila Pa 1976). 2003 Jan 1;28(1):74-8. doi: 10.1097/00007632-200301010-00017. PMID 12544960
- [Background] Yagci G, Yakut Y. Core stabilization exercises versus scoliosis-specific exercises in moderate idiopathic scoliosis treatment. Prosthet Orthot Int. 2019 Jun;43(3):301-308. doi: 10.1177/0309364618820144. Epub 2019 Jan 10. PMID 30628526